CLINICAL TRIAL: NCT05148871
Title: A Phase 2b Study to Assess the Effect of Dose Interval on the Effectiveness of a Protein-based Covid-19 Vaccine (Spikogen® Vaccine)
Brief Title: Australian Phase 2b Study to Assess Effect of Dose Interval on Spikogen Covid-19 Vaccine
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute (Other); Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C19-P2/3B
Record Dates: First submitted 2021-11-27; First posted 2021-12-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: covid-19; SARS-CoV-2; coronavirus; vaccine; adjuvant; Advax
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Intervention Model Description: Subjects will be randomised into 4 groups, where the only difference will be the time between vaccine doses (3, 4, 5 or 6 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 week arm (Active Comparator): Subjects will receive two doses of vaccine 3 weeks apart
  Interventions: Biological: Spikogen/Covax-19
- 4 week arm (Active Comparator): Subjects will receive two doses of vaccine 4 weeks apart
  Interventions: Biological: Spikogen/Covax-19
- 5 week arm (Active Comparator): Subjects will receive two doses of vaccine 5 weeks apart
  Interventions: Biological: Spikogen/Covax-19
- 6 week arm (Active Comparator): Subjects will receive two doses of vaccine 6 weeks apart
  Interventions: Biological: Spikogen/Covax-19

INTERVENTIONS:
Biological: Spikogen/Covax-19 — Spikogen/Covax-19 is a recombinant spike protein vaccine formulated with Advax-CpG55.2 adjuvant

SUMMARY:
A study to assess the effect of varying the time interval between doses on the immunogenicity of an adjuvanted recombinant spike protein Covid-19 vaccine (Spikogen/Covax-19)

DETAILED DESCRIPTION:
The SARS-CoV-2 outbreak has caused millions of deaths globally. It has a particularly high mortality rate in elderly people and those with chronic disease where mortality rates can be as high as 20-30%. SARS-COV-2 vaccines remain a key priority to help fight the current pandemic and prepare for future coronavirus outbreaks. COVID-19 vaccines have potential to prevent symptomatic infections and may help reduce virus transmission. Covax-19/Spikogen is the first full length recombinant spike protein vaccine in the world to receive emergency use authorisation after it was shown in Phase 3 trials to be 60-65% effective at preventing symptomatic infection with the delta variant. It has been reported for other Covid-19 vaccines that a longer dose interval between first and second doses may further increase vaccine immunogenicity and protection. As a 3-week dose interval was tested in the clinical trials that supported Spikogen's authorisation, it will be beneficial to test whether a longer dose interval than 3 weeks may have a favourable effect on vaccine immunogenicity and thereby protection.

SARS-CoV-2 is an enveloped, single positive-stranded RNA virus, with one genome encoding a non-structural replicase polyprotein and structural proteins including spike (S), envelope (E), membrane (M) and nucleocapsid (N) proteins. Neutralizing antibodies are directed against the S protein receptor binding domain (RBD). T cells directed against the S protein may also play a role in protection and virus clearance.

Spikogen, also known under the Covax-19 tradename in Australia, is based on recombinant SARS-COV-2 spike protein manufactured in insect cells that is formulated with a combination adjuvant known as Advax-CpG55.2. Insect cell expression of recombinant protein is a well-established vaccine manufacturing approach. The purified recombinant protein is formulated with Advax-CpG55.2 adjuvant to ensure a sufficiently robust immune response enabling the vaccine to produce protective levels of immunity. Advax-CpG55.2 has two components, one a natural plant sugar called inulin and the second a short synthetic polymer made up of oligonucleotides, known as CpG55.2. Advax-CpG adjuvant has been used in multiple human clinical trials of influenza and Covid-19 vaccines and has been found to be safe and well tolerated, just causing a mild increase in local injection site soreness when compared to a saline injection.

Spikogen vaccine is designed to protect against SARS-CoV-2 infection by generation of antibodies and memory cells against the spike protein. It has been shown to provide protection against SARS-CoV-2 virus infection in hamster, ferret and monkey models. In the hamster model it was shown to provide protection against the original Wuhan strain as well as against the more recent beta and Delta variant strains. In preclinical studies it was well tolerated and caused no major adverse reactions. Following successful completion of a Phase 2 trial in 400 adult participants that confirmed its safety and immunogenicity, a Phase 3 clinical trial was undertaken in Iran involving 16,876 participants randomised 3:1 to receive active vaccine or placebo using two intramuscular doses administered 3 weeks apart. Spikogen vaccine successfully met its prespecified primary efficacy endpoint established by the Iranian FDA, namely demonstration of >60% protection against symptomatic PCR-confirmed infection. On this basis of efficacy shown in the Phase 3 trial, Spikogen received emergency use authorisation by the Iranian FDA in October 2021, making it the first such vaccine in the world to receive authorisation. Since its authorisation more than 1 million doses of Spikogen vaccine have been safely delivered.

It is now planned to undertake a clinical trial in Australia to determine, based on measurement of anti-spike antibody levels, the optimal time between the two doses when the vaccine is used as a primary immunisation regimen in vaccine-naive individuals.

Rationale for schedule of administration The aim is to determine the best dose interval for a course of 2 doses in vaccine naïve individuals. This trial will administer two doses of vaccine to vaccine-naïve individuals at variable intervals (3, 4, 5 or 6 weeks) to assess the effect of timing of the second vaccine dose on anti-spike protein antibody production.

Rationale for selection of doses In the Phase 3 clinical trial, two 25 ug doses of vaccine given 3 weeks apart provided 60-65% protection against symptomatic SARS-CoV-2 infection with the delta strain. This trial will test the same dose of the authorised vaccine as used in the pivotal Phase 3 trial but just with a varying time window between the two doses.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study procedures.
* No history of previous Covid-19 vaccinations
* Women of childbearing potential must use an acceptable contraception method from at least 28 days before study vaccination until 14 days after last study vaccination.
* Understand and comply with planned study procedures and be available for all study visits.

Exclusion Criteria:

* Have a history of severe systemic reactions (anaphylaxis, breathing difficulties, severe rash) following previous immunization with licensed or unlicensed vaccines.
* Received an experimental agent within 30 days prior to the study vaccination or expect to receive another experimental agent during the trial-reporting period.
* Intend to receive another Covid-19 vaccine during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2024-10-06 (Estimated)

PRIMARY OUTCOMES:
Spike antibody immunogenicity | 3 weeks post second vaccine dose
  Serum geometric mean titers of anti-spike protein antibody levels
Spike antibody seroconversion | 3 weeks post second vaccine dose
  Proportion of each group seroconverting to spike protein antibody positiivity
SARS-CoV-2 protection | Accrual of events starting 2 weeks post second vaccine dose
  Confirmed Covid-19 infections

SECONDARY OUTCOMES:
Spike antibody durability | 6 months post-second vaccine dose
  Serum geometric mean titers of anti-spike protein antibodies
Spike antibody seropositive persistence | 6 months post-second vaccine dose
  Proportion of each group remaining seropositive for anti-spike antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, MD, PhD, Principal Investigator — ARASMI
Locations (1):
- ARASMI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li L, Honda-Okubo Y, Huang Y, Jang H, Carlock MA, Baldwin J, Piplani S, Bebin-Blackwell AG, Forgacs D, Sakamoto K, Stella A, Turville S, Chataway T, Colella A, Triccas J, Ross TM, Petrovsky N. Immunisation of ferrets and mice with recombinant SARS-CoV-2 spike protein formulated with Advax-SM adjuvant protects against COVID-19 infection. Vaccine. 2021 Sep 24;39(40):5940-5953. doi: 10.1016/j.vaccine.2021.07.087. Epub 2021 Aug 3. PMID 34420786
- [Background] Tabarsi P, Anjidani N, Shahpari R, Mardani M, Sabzvari A, Yazdani B, Roshanzamir K, Bayatani B, Taheri A, Petrovsky N, Li L, Barati S. Safety and immunogenicity of SpikoGen(R), an Advax-CpG55.2-adjuvanted SARS-CoV-2 spike protein vaccine: a phase 2 randomized placebo-controlled trial in both seropositive and seronegative populations. Clin Microbiol Infect. 2022 Sep;28(9):1263-1271. doi: 10.1016/j.cmi.2022.04.004. Epub 2022 Apr 15. PMID 35436611
- [Background] Li L, Honda-Okubo Y, Baldwin J, Bowen R, Bielefeldt-Ohmann H, Petrovsky N. Covax-19/Spikogen(R) vaccine based on recombinant spike protein extracellular domain with Advax-CpG55.2 adjuvant provides single dose protection against SARS-CoV-2 infection in hamsters. Vaccine. 2022 May 20;40(23):3182-3192. doi: 10.1016/j.vaccine.2022.04.041. Epub 2022 Apr 18. PMID 35465982